CLINICAL TRIAL: NCT06885879
Title: Impact of Radiotherapy on the Dynamic Changes of Circulating Cell-free DNA in Patients With Hepatocellular Carcinoma
Brief Title: Impact of Radiotherapy on ctDNA in Patients With Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Landon Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: TRA025
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temporal change of fragmentomics of Circulating tumour DNA investigation
  Interventions: Radiation: Temporal change of fragmentomics of Circulating tumour DNA undergoing Stereotactic Body Radiation Therapy investigation

INTERVENTIONS:
Radiation: Temporal change of fragmentomics of Circulating tumour DNA undergoing Stereotactic Body Radiation Therapy investigation — Patients will have blood taking for Circulating tumour DNA (ctDNA) (20cc each) at Week 0 (before radiotherapy), Week 1 (during radiotherapy), Week 2 (after radiotherapy), Week 12 and Week 24.
  Radiological assessment will be performed before radiotherapy, Week 12 (approximately 3 months post treatment) and Week 24-26 (approximately 6 months post treatment).

SUMMARY:
Radiotherapy is increasingly being used in the management of hepatocellular carcinoma (HCC) as a standalone treatment, or in combination with systemic therapy. Stereotactic Body Radiation Therapy (SBRT) causes cell death directly (via double-stranded breaks) and indirectly (via vascular bed damage or promotion of antitumour immunity). Unfortunately, the effect of cell death is not immediate and takes time. As a result, the typical arterial phase hyperenhancement on imaging may persist up to 12 months after radiotherapy, and it is not necessarily suggestive of presence of viable tumours. Therefore, there is no consensus on ideal timing of response assessment following radiotherapy to HCC. Therefore, a blood-based biomarker which can be done frequently and monitored dynamically, could be preferred for response assessment after radiotherapy. Circulating tumour DNA (ctDNA) is an emerging and promising biomarker in cancer management, which has been shown useful in cancer screening, guiding treatment, and informing prognosis. Currently, most of the clinical applications of ctDNA revolve around either the presence of ctDNA, or the genomic changes associated with these molecules. Biological properties of ctDNA such as fragment length, jaggedness of fragments, or epigenetic changes may provide additional information related to the tumour characteristics and its sensitivity to anti-cancer treatments. These biological properties of ctDNA are relatively unexplored in the context of radiotherapy. It is unknown whether these properties can be utilized for monitoring treatment response. We therefore propose to study the biological properties of ctDNA in relation to HCC patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance 0 to 1
* Confirmed diagnosis of Hepatocellular carcinoma (HCC)
* Tumour size ≥ 3cm
* Patients planning on undergoing Stereotactic Body Radiation Therapy (SBRT) for HCC
* Prior radiofrequency ablation at a different site, or prior surgery are eligible
* Child-Pugh A liver function
* Life expectancy longer than 12 weeks
* At least one measurable treatment lesion according to RECIST 1.1
* Written informed consent must be obtained prior to any study related procedures
* Adequate haematological function (Hemoglobin ≥ 8.5g/dL; Platelet Count ≥ 75x109/L; Antenatal Care ≥ 1.5x109/L; international normalised ratio ≤ 1.5)
* Adequate hepatic function (albumin ≥ 28g/l; Bilirubin ≤ 1.5xULN; Alanine transaminase < 5 times upper limit normal)
* Adequate renal function (serum creatinine ≤ 1.5 times the upper limit of normal range; Sodium ≥ 130mmol/L; Potassium ≥ 3.0mmol/L)
* Able to read, understand and provide written consent

Exclusion Criteria:

* Histology shows sarcomatoid HCC, fibrolamellar HCC, mixed cholangiocarcinoma-hepatocellular carcinoma
* Presence of other malignancy than HCC within 5 years from diagnosis of HCC
* Prior Transarterial chemoembolization (TACE) within 3 months
* Previous radiotherapy to the abdomen
* Previous yttrium-90 chemoembolization
* Repetitive history of non-healing wounds or ulcers within 2 months of inclusion
* Pregnant or lactating females at any time during the study
* Active autoimmune disease requiring systemic therapy in the past 2 years
* Diagnosis of immunodeficiency (including Human Immunodeficiency Viruses)
* Patients with coagulopathy or on anticoagulant will be excluded from liver biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the temporal changes of the biological properties of Circulating tumour DNA, including its relative percentage, fragment size, and end-motif fragment pattern for patients undergoing radiotherapy to Hepatocellular carcinoma. | 2 years

SECONDARY OUTCOMES:
To correlate the change in biological properties with response (by RECIST 1.1), survival (e.g. progression-free survival), and toxicities | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong